CLINICAL TRIAL: NCT03586492
Title: SPECT Myocardial Perfusion Reserve Using a Cadmium Zinc Telluride (CZT) Camera in Cardiovascular Risk Stratification and Ischemia
Brief Title: Coronary Flow Reserve (CFR) in Cardiovascular Risk Stratification
Acronym: CFR-OR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2018-05
Record Dates: First submitted 2018-07-03; First posted 2018-07-13 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Ischemia, Myocardial; Ischemic Heart Disease
Keywords: CFR; SPECT; CZT; Coronary; Calcium score; Scintigraphy; Myocardial perfusion
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with myocardial ischemia (Other)
  Interventions: Diagnostic Test: CZT SPECT acquisition

INTERVENTIONS:
Diagnostic Test: CZT SPECT acquisition — CZT SPECT acquisition, with dynamic stress and rest acquisitions to calculate CFR If pathological, coronarography with FFR measurement if necessary In case of intermediate coronary stenosis with medical treatment, SPECT CFR evaluation after one year of treatment

SUMMARY:
CFR has been studied for few years using 82 Rubidium PET (positron emission tomography) /CT. CFR has shown to be correlated with cardiovascular events occurring in the 10 following years. CFR also helps to identify multivessel coronary disease. Few studies have shown the possibility to calculate CFR during myocardial perfusion SPECT on new ultrafast CZT cameras.

DETAILED DESCRIPTION:
Evaluate the contribution of CZT SPECT CFR in cardiovascular risk stratification: correlation with clinical scores, with calcium score, and when pathological with coronarography findings especially fractional flow reserve (FFR).

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for myocardial ischemia screening

Exclusion Criteria:

* Patient already suffering from coronary disease with angioplasty, bypass surgery or myocardial infarction.
* Contraindications related to the stress test:

Acute Coronary Syndrome <5 days Unstable angina Stenosis of left main artery untreated Uncontrolled severe rhythm disorders Uncontrolled heart failure

* Contraindications to dipyridamole and regadenoson:

Hypotension (systolic <90mmHg) Severe pulmonary arterial hypertension Bradycardia <40 beats / minute Sinusal Dysfunction and 2nd or 3rd degree Atrioventricular block Decompensated Heart Failure with Ejection Fraction <25% Stenosis of supra-aortic trunks unilateral> 70% or bilateral> 50% Dipyridamole and regadenoson allergy

* Patients with pacemaker, or who have had valvular surgery,
* Well-known dilated cardiopathy
* Pregnant or breastfeeding women,
* Minor people
* Persons under guardianship or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Regional and global CFR | Day 0
  Regional and global CFR calculated from CZT SPECT myocardial perfusion: correlation with clinical score and calcium score

SECONDARY OUTCOMES:
FFR Regional CFR after one year of medical treatment | Up to one year
  FFR measured during coronarography if there is an intermediate stenosis Regional CFR if there is an intermediate coronary stenosis with medical treatment, after one year of treatment, calculated during a new SPECT CZT exam

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu BAILLY, Dr, Principal Investigator — CHR d'Orléans
Locations (2):
- France (2):
  - CHR d'Orleans, Orléans
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agatston AS, Janowitz WR, Hildner FJ, Zusmer NR, Viamonte M Jr, Detrano R. Quantification of coronary artery calcium using ultrafast computed tomography. J Am Coll Cardiol. 1990 Mar 15;15(4):827-32. doi: 10.1016/0735-1097(90)90282-t. PMID 2407762
- [Background] Agostini D, Roule V, Nganoa C, Roth N, Baavour R, Parienti JJ, Beygui F, Manrique A. First validation of myocardial flow reserve assessed by dynamic 99mTc-sestamibi CZT-SPECT camera: head to head comparison with 15O-water PET and fractional flow reserve in patients with suspected coronary artery disease. The WATERDAY study. Eur J Nucl Med Mol Imaging. 2018 Jul;45(7):1079-1090. doi: 10.1007/s00259-018-3958-7. Epub 2018 Mar 1. PMID 29497801
- [Background] Assante R, Zampella E, Arumugam P, Acampa W, Imbriaco M, Tout D, Petretta M, Tonge C, Cuocolo A. Quantitative relationship between coronary artery calcium and myocardial blood flow by hybrid rubidium-82 PET/CT imaging in patients with suspected coronary artery disease. J Nucl Cardiol. 2017 Apr;24(2):494-501. doi: 10.1007/s12350-015-0359-1. Epub 2016 Jan 15. PMID 26780529
- [Background] Ben Bouallegue F, Roubille F, Lattuca B, Cung TT, Macia JC, Gervasoni R, Leclercq F, Mariano-Goulart D. SPECT Myocardial Perfusion Reserve in Patients with Multivessel Coronary Disease: Correlation with Angiographic Findings and Invasive Fractional Flow Reserve Measurements. J Nucl Med. 2015 Nov;56(11):1712-7. doi: 10.2967/jnumed.114.143164. Epub 2015 Sep 3. PMID 26338893